CLINICAL TRIAL: NCT06570798
Title: A Phase 2a, Open Label, Multicenter, Platform Trial to Assess the Safety, Tolerability, and Efficacy of Inebilizumab and Blinatumomab in Subjects With Autoimmune Diseases
Brief Title: A Phase 2a Master Protocol Assessing Inebilizumab and Blinatumomab in Autoimmune Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240033; 2024-514382-19 (EudraCT Number)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus; Active Refractory Rheumatoid Arthritis
Keywords: Systemic lupus erythematosus; Inebilizumab; Blinatumomab; Active refractory rheumatoid arthritis; Rheumatoid arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid | interventions — inebilizumab; blinatumomab

STUDY DESIGN:
Intervention Model Description: Subprotocol A: Sequential study model Subprotocol B: Sequential study model Subprotocol C: Sequential study model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Subprotocol A: Inebilizumab 3 Doses (Experimental): Participants will receive 3 doses of inebilizumab administered via an intravenous (IV) infusion.
  Interventions: Drug: Inebilizumab
- Subprotocol A: Inebilizumab 4 Doses (Experimental): Participants will receive 4 doses of inebilizumab administered via an IV infusion.
  Interventions: Drug: Inebilizumab
- Subprotocol B: Blinatumomab Low-dose (Experimental): Participants will receive blinatumomab low-dose administered via SC injection.
  Interventions: Drug: Blinatumomab
- Subprotocol B: Blinatumomab Medium-dose (Experimental): Participants will receive blinatumomab medium-dose administered via SC injection.
  Interventions: Drug: Blinatumomab
- Subprotocol B: Blinatumomab High-dose (Experimental): Participants will receive blinatumomab high-dose administered via SC injection.
  Interventions: Drug: Blinatumomab
- Subprotocol C: Blinatumomab Low-dose (Experimental): Participants will receive blinatumomab low-dose administered via SC injection.
  Interventions: Drug: Blinatumomab
- Subprotocol C: Blinatumomab Medium-dose (Experimental): Participants will receive blinatumomab medium-dose administered via SC injection.
  Interventions: Drug: Blinatumomab
- Subprotocol C: Blinatumomab High-dose (Experimental): Participants will receive blinatumomab high-dose administered via SC injection.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Inebilizumab — Intravenous (IV) Infusion
  Other Names: Uplizna®
  Arms: Subprotocol A: Inebilizumab 3 Doses; Subprotocol A: Inebilizumab 4 Doses
Drug: Blinatumomab — SC Injection
  Arms: Subprotocol B: Blinatumomab High-dose; Subprotocol B: Blinatumomab Low-dose; Subprotocol B: Blinatumomab Medium-dose; Subprotocol C: Blinatumomab High-dose; Subprotocol C: Blinatumomab Low-dose; Subprotocol C: Blinatumomab Medium-dose

SUMMARY:
The main objective is to assess the safety and tolerability of inebilizumab in adult participants with active and refractory systemic lupus erythematosus (SLE) with nephritis (Subprotocol A) and to assess the safety and tolerability of subcutaneous (SC) blinatumomab in adult participants with active and refractory SLE with and without nephritis (Subprotocol B) and in adult participants with active refractory rheumatoid arthritis (RA) (Subprotocol C).

ELIGIBILITY:
Inclusion Criteria:

* Subprotocol A and B: Diagnosis of SLE according to 2019 European League Against Rheumatism and the American College of Rheumatology (ACR) classification criteria.
* Subprotocol A and B: Participant must be positive for at least one of the following autoantibodies at screening (performed by central laboratory) or through documented history:

  1. Antinuclear antibodies (ANA) ≥ 1:80
  2. Anti-double stranded deoxyribonucleic acid (anti-dsDNA) antibodies elevated to above normal range (ie, positive results)
  3. Anti-Smith antibodies elevated to above normal (ie, positive results).
* Subprotocol A and B (with LN): Active, biopsy-proven, proliferative LN demonstrating class III or class IV with or without co-existing features of Class V LN (or pure Class V LN for Subprotocol B only) according to 2018 International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria. The local biopsy report will be used.
* Subprotocol A and B (with LN): Systemic Lupus Erythematosus Disease Activity Index 2K ≥ 6.
* Subprotocol A and B (with LN): Inadequate response, loss of response or intolerance to at least 1 therapy (Subprotocol A) or 2 immunosuppressive therapies (Subprotocol B with LN) at the maximally tolerated doses as recommended by the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines (KDIGO, 2024). Inadequate response is defined as: UPCR ≥ 1.0 mg/mg.
* Subprotocol B (SLE without nephritis): Systemic Lupus Erythematosus Disease Activity Index 2K ≥ 6.
* Subprotocol B (SLE without nephritis): Refractory SLE participants with inadequate response to multiple therapies (excluding hydroxychloroquine or corticosteroids) and have failed either a biologic agent or cyclophosphamide.
* Subprotocol A and B: If receiving any of the following medications, participants must be on these doses prior to day 1:

  1. Prednisone dose ≤ 20 mg/day (or its equivalent in other corticosteroid forms) and at a stable dose for 5 days
  2. Hydroxychloroquine dose ≤ 400 mg/day and at a stable dose for 4 weeks. Other equivalent antimalarials (chloroquine, quinacrine) are also accepted at a stable dose for 4 weeks.
  3. MMF dose ≤ 3 g/day or MPA dose ≤ 2160 mg/day and at a stable dose for 2 weeks.
  4. AZA dose ≤ 2 mg/kg/day and at a stable dose for 2 weeks.
* Subprotocol C: Diagnosis of RA according to the 2010 ACR/ European Alliance of Associations for Rheumatology (EULAR) classification criteria.
* Subprotocol C: Moderate to severe disease activity as defined by DAS28-CRP > 3.2 with ≥ 3 swollen joints and ≥ 3 tender joints (based on 28 joint counts) at screening.
* Subprotocol C: Refractory disease defined as:
* Moderate to severe active disease despite having received treatment with:

  1. at least 1 conventional synthetic disease-modifying antirheumatic drug (csDMARD), AND
  2. at least 2 biologic disease-modifying antirheumatic drugs (bDMARDs) of different mechanisms of action OR 1 bDMARD and at least 1 targeted synthetic disease-modifying antirheumatic drugs (tsDMARD).
* Inadequate response or intolerance to csDMARDs, bDMARDs, and tsDMARDs should be defined as:

  1. Participant having active disease despite a minimum of 12 weeks of treatment with a csDMARD, bDMARD, or tsDMARD.
  2. Intolerance to treatment as defined by participant having experienced an adverse effect from treatment with a csDMARD, bDMARD, or tsDMARD.

Exclusion Criteria:

* Subprotocol A and B: Estimated glomerular filtration rate (eGFR) of < 30 mL per minute per 1.73 m^2 of body surface area (calculated using the Modification of Diet in Renal Disease [MDRD] formula, with screening laboratory results for serum creatinine value).
* Subprotocol A and B: Significant likely irreversible organ damage related to SLE (eg, end-stage renal disease [ESRD]).
* Subprotocol A and B: Any acute, severe lupus related flare during screening that needs immediate treatment.
* Subprotocol A and B: A previous kidney transplant or planned transplant within study treatment period.
* Subprotocol A and B: History of or current renal diseases (other than LN) that in the opinion of the investigator could interfere with the LN assessment and confound the disease activity assessment (eg, diabetic nephropathy).
* Subprotocol A: Renal biopsy showing pure class V.
* Subprotocol C: Prior history of current inflammatory joint disease other than RA including but not limited to systemic lupus erythematosus, mixed connective tissue disorder, scleroderma, polymyositis, or significant systemic involvement secondary to RA (eg, vasculitis, pulmonary fibrosis, or Felty's syndrome).
* Subprotocol C: Functional Class IV as defined by the ACR classification of functional status in RA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-06-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 to Week 52
Number of Participants Who Experience a Serious TEAE | Day 1 to Week 52

SECONDARY OUTCOMES:
Subprotocol A and B: Number of Participants With Complete Renal Response (CRR) | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Number of Participants With Partial Renal Response (PRR) | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Number of Participants With Remission in SLE as Defined by Definition of Remission in SLE (DORIS) | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Number of Participants With a Lupus Low Disease Activity State (LLDAS) | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Change From Baseline in SLE Activity Index-2000 (SLEDAI-2K) Score | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Percent Change From Baseline in SLEDAI-2K Score | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Change From Baseline in 24-hour UPCR | Week 12, Week 26, Week 38, and Week 52
Subprotocol A and B: Percent Change From Baseline in 24-hour UPCR | Week 12, Week 26, Week 38, and Week 52
Subprotocol A: Maximum Concentration (Cmax) of Inebilizumab | Day 1 to Week 52
Subprotocol A: Time to Cmax (tmax) of Inebilizumab | Day 1 to Week 52
Subprotocol A: Area Under the Concentration-time Curve (AUC) of Inebilizumab | Day 1 to Week 52
Subprotocol B and C: Cmax of Blinatumomab | Day 1 to Week 12
Subprotocol B and C: tmax of Blinatumomab | Day 1 to Week 12
Subprotocol B and C: AUC of Blinatumomab | Day 1 to Week 12
Subprotocol A: Number of Participants With Anti-inebilizumab Antibody Formation | Day 1 to Week 52
Subprotocol B and C: Number of Participants With Anti-blinatumomab Antibody Formation | Day 1 to Week 52
Subprotocol C: Percentage of participants achieving Disease Activity Score-28 Joint C-Reactive Protein (DAS28-CRP) < 2.6 | Week 12 and Week 26
Subprotocol C: Percentage of participants achieving Clinical Disease Activity Index (CDAI) ≤ 2.8 | Week 12 and Week 26
Subprotocol C: Percentage of participants achieving Simplified Disease Activity Index (SDAI) ≤ 3.3 | Week 12 and Week 26
Subprotocol C: Percentage of participants achieving American College of Rheumatology (ACR)20 response | Week 12 and Week 26
Subprotocol C: Percentage of participants achieving ACR50 response | Week 12 and Week 26
Subprotocol C: Percentage of participants achieving ACR70 response | Week 12 and Week 26

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (45):
- United States (11):
  - HonorHealth Research and Innovation Institute, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Vida Research Center, Hialeah, Florida
  - Homestead Associates In Research Inc, Homestead, Florida
  - Vitaly Clinical Research, Miami, Florida
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Prolato Clinical Research Center, Houston, Texas
- Linear Clinical Research Limited, Perth, Western Australia, Australia
- Belgium (4):
  - Cliniques Universtaire Saint Luc Universite Catholique de Louvain, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- France (12):
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Lyon- Hopital Edouard Herriot, Lyon
  - Centre Hospitalier Universitaire de Lyon - Hopital Edouard Herriot, Lyon Cédex 3
  - Hopital de la Conception, Marseille
  - Hopital Cochin, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Strasbourg - Hopital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Purpan, Toulouse
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
- Germany (4):
  - Krankenhaus Porz am Rhein gGmbH, Cologne
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der LMU Muenchen, München
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Ospedale San Giovanni Bosco, Torino
- Portugal (3):
  - Unidade Local de Saude de Lisboa Ocidental, EPE - Hospital Santa Cruz, Carnaxide
  - Unidade Local de Saude de Sao Jose, EPE - Hospital Curry Cabral, Vila Franca de Xira
  - Unidade Local de Saude de Gaia-Espinho, EPE, Vila Nova de Gaia
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Addenbrookes Hospital, Cambridge
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com